CLINICAL TRIAL: NCT02703571
Title: A Phase I/II Study of Safety and Efficacy of Ribociclib (LEE011) in Combination With Trametinib (TMT212) in Patients With Metastatic or Advanced Solid Tumors
Brief Title: Study of Safety and Efficacy of Ribociclib and Trametinib in Patients With Metastatic or Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMT212X2106; 2015-005019-34 (EudraCT Number)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors for Phase Ib; Pancreatic Cancer for Phase II; Colorectal Cancer for Phase II
Keywords: Trametinib; Ribociclib; LEE011; TMT212; advanced solid tumors; pancreatic cancer; KRAS-mutant colorectal cancer; colorectal cancer; advanced pancreatic cancer; metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms | interventions — ribociclib; trametinib

STUDY DESIGN:
Intervention Model Description: single group for phase 1b parallel group for phase 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advanced or metastatic solid tumors (Experimental): Patients in the Phase I portion of the study who have advanced or metastatic solid tumors
  Interventions: Drug: ribociclib; Drug: Trametinib

INTERVENTIONS:
Drug: ribociclib — Combination treatment with LEE and TMT
  Other Names: LEE011
Drug: Trametinib — Combination treatment with LEE and TMT
  Other Names: TMT212

SUMMARY:
Phase Ib dose escalation in advanced solid tumors to identify dose for Phase II dose expansion in advanced or metastatic pancreatic cancer and KRAS-mutant colorectal cancer. Open-label, nonrandomized.

DETAILED DESCRIPTION:
Upon careful review of all available efficacy and safety data from the study phase Ib part, Novartis decided to not start the study phase II part.

This decision was in no means triggered by an unfavorable safety profile of the combination. The observed safety profile of the combination represents contributions of the individual safety profile of trametinib and ribociclib.

No new safety signals were observed.

The study was closed early in line with protocol Section 4.4.

ELIGIBILITY:
Inclusion Criteria (All):

* Written informed consent must
* Patient has histologically and/or cytologically confirmed malignancies:

Phase I:

• Patients with advanced or metastatic solid tumors who have failed at least one prior line of systemic antineoplastic therapy in the advanced setting without a standard of care treatment option available;

Phase II:

* Advanced or metastatic pancreatic adenocarcinoma who have failed at least one prior systemic antineoplastic therapies in the advanced setting
* Advanced or metastatic KRAS-mutant CRC who have failed at least two prior systemic antineoplastic therapies in the advanced setting without a standard of care treatment option available. Testing for KRAS mutation in patients with CRC using locally approved diagnostic kit will be used for eligibility.
* Phase II only: patient must have measurable disease
* Patient has an ECOG performance status 0 or 1.
* Patient has adequate bone marrow and organ function
* Patient must have specified laboratory values within normal limits or corrected to within normal limits with supplements before the first dose of study medication on Cycle 1 Day 1:
* Standard 12-lead ECG values defined

Exclusion Criteria:

Phase II only:

• Patient has received prior treatment with a MEK inhibitor or a CDK4/6 inhibitor.

Phase I and Phase II:

* Patient with a known hypersensitivity to the study drugs or any of the excipients of ribociclib or trametinib.
* Patient is concurrently using other anti-cancer therapy.
* Patient has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to Cycle 1 Day 1
* Patient has received local therapy to liver ≤ 3 months of C1D1
* History of liver disease as follow:
* Cirrhosis
* Autoimmune hepatitis
* Active viral hepatitis
* Portal hypertension
* Drug induced liver steatosis
* Prior systemic anti-cancer treatment within 28 days prior to Cycle 1 Day 1
* Prior therapy with anthracyclines at cumulative doses of 450 mg/ m2 or more for doxorubicin or 900 mg/m2 or more for epirubicin.
* Patient is currently receiving warfarin or other coumadin derived anti-coagulant
* Patient has a history of deep venin thrombosis or pulmonary embolism within 6 months of screening.
* Patient has a concurrent malignancy or malignancy within 3 years prior to Cycle 1 Day 1, with the exception of adequately treated basal or squamous cell carcinoma or curatively resected cervical cancer.
* Patients with central nervous system (CNS) involvement
* Patient has impairment of GI function or GI disease that may significantly alter the absorption of the study drugs
* History of interstitial lung disease or pneumonitis.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality
* Patient is currently receiving any strong inducers or inhibitors of CYP3A4/5 and/or Substances that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5 and cannot be discontinued 7 days prior to Cycle 1 Day 1:
* Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.
* History of retinal vein occlusion (RVO)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | 21-day cycle one of treatment
  Phase Ib part:
  The primary variable is the incidence of DLTs during the first 21 days of therapy. Estimation of the MTD of the combination treatment will be based upon the estimation of the probability of DLT during the first 21 days of therapy for patients in the DDS.
Objective Response Rate (ORR) | Until progression of disease up to 1 year
  Phase II part:
  The primary variable used to evaluate the efficacy of the ribociclib and trametinib combination is the ORR, defined as the proportion of patients with a best overall confirmed CR or PR, as assessed per RECIST 1.1 by investigator assessment.

SECONDARY OUTCOMES:
Duration of response (DOR) | Until progression of disease up to 1 year
  Phase II part:
  Among patients with a confirmed response (PR or CR) per RECIST 1.1, DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause. The distribution function of DOR will be estimated using the Kaplan-Meier method. The median DOR along with 95% CI will be presented by treatment arm.
Time to response | Until progression of disease up to 1 year
  Phase II part:
  Time to overall response of CR or PR (TTR) is defined as the time from start of study drug to first documented response (CR or PR, which must be confirmed subsequently) for patients with a confirmed CR or PR. TTR will be summarized by treatment arm, using descriptive statistics.
Disease control rate | Until progression of disease up to 1 year
  Phase II part:
  Disease control rate (DCR) is defined as the proportion of patients with best overall response of CR, PR, or SD per RECIST 1.1. DCR will be estimated and the binomial exact 95% CI will be provided by arm.
Progression disease rate | Until progression of disease up to 1 year
  Phase Ib part:
  Progression disease rate defined as the proportion of patients with a progression disease as assessed per RECIST 1.1 by investigator assessment.
Progression free survival | Until progression of disease up to 1 year
  Phase Ib and phase II parts:
  Progression-free survival (PFS) is defined as the time from the date of the first dose of study drug to the date of first documented disease progression per RECIST 1.1 or death due to any cause.
overall survival | Until death up to 1 year
  Phase Ib and phase II parts:
  Overall survival (OS) is defined as the time from the date of first dose of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (6):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami Sylvester Comp Cancer Ctr, Miami, Florida
  - Dana Farber Cancer Center, Boston, Massachusetts
  - UT MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Ulm
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Results for CTMT212X2106 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17721